CLINICAL TRIAL: NCT06278584
Title: The iLux and Mechanical Meibomian Gland Expression for the Treatment of Moderate and Severe Meibomian Gland Dysfunction.
Brief Title: iLux Treatment for Meibomian Gland Dysfunction
Acronym: MGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica de Oftalmología de Cali S.A (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020001-00
Record Dates: First submitted 2024-02-06; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Meibomian Gland Dysfunction; Eyes Dry Chronic
Keywords: Meibomian Gland Dysfunction; ILux®; ocular surface; dry eye
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- iLUX Treatment System (Active Comparator): The eyelid tissue is warmed by light energy produced by LEDs in the Instrument and transmitted through the precise Outer Pad. The Inner Pad and Eye Shield block light transmission directly into the eye during a treatment temperature sensor and measure the inner and outer eyelid temperatures to maintain a meibum melt temperature of 38-42°C.
  Interventions: Device: iLUX Treatment System
- Mechanical Meibomian Gland Expression (Active Comparator): 1. Local heat using an electrical warming mask for 5 minutes.
  2. Using a standardized device (Arita Meibomian Gland Compressor, Katena) to apply a standard force to individual glands
  Interventions: Device: iLUX Treatment System

INTERVENTIONS:
Device: iLUX Treatment System — Local heat using an electrical warming mask for 5 minutes.
  Other Names: Mechanical Meibomian Gland Expression

SUMMARY:
Summary:

Purpose: To compare the safety and efficacy of eyelid treatment with the ILux®-MGD Treatment System in one session versus five sessions of mechanical meibomian gland expression (MMGE) in patients with moderate to severe meibomian gland dysfunction (MGD).

Methods: Prospective, randomized, open-label, controlled clinical trial comparing one session of the ILux® MGD Treatment System versus five sessions of MMGE in both eyes of 130 patients aged ≥18 years with OSDI scores ≥13, total MGS of 15 in the lower lid of each eye and NI-TBUT <10 s, who were randomized 1:1 to ILux® or MMGE.

DETAILED DESCRIPTION:
Meibomian glands (MG) are responsible for the secretion of lipids (meibum) into the ocular surface and have a protective role for tear film against evaporation1-4; therefore, Meibomian Gland Dysfunction (MGD) is associated with evaporative dry eye (EDE). Hyperkeratinization and hyperviscosity occur in dysfunctions with low MG expressibility, low meibum quality and eyelid margin inflammation. Finally, atrophy and dropout of MGs in some cases could appear MGD is a prevalent dry eye disorder (DED) with an estimated prevalence range between 3.5% and 70%1,10-13, it constitutes the primary underlying pathology within the EDE subtype. On top of this, MGD is chronic and progressive, so it is imperative to identify clinical approaches that can effectively target this underlying condition.

Treatment of MGD often involves artificial lubricants, topical lipid supplements, lid hygiene, warm compression or heat application, supplement omega-3, topical and systemic antibiotics against Demodex mite infestation, and steroids.

Mechanical management involves debridement-scaling of the line of Marx and lowers lid margin21, and other methods for mechanical manual expression in alignment with the concept that optimal treatment of MGD requires the employment of some forms of evacuating MGs contents.

Eyelid thermal pulsation devices combine the application of heat at the appropriate temperature to the palpebral surface with simultaneous compression of the glands to evacuate their contents, and have been shown to improve signs and symptoms over 12 months in cases of severe meibomian obstruction.

More recently, the ILux® MGD Treatment System (Alcon, FortWorth, TX, USA) is an eyelid thermal pulsation system that includes a single-use patient interface device and a portable battery-powered instrument that simultaneously applies localized heat and compression to treat MGD and showed significant improvements in MG function between one and four weeks.

Prior to the introduction of vectored thermal pulsation therapies, the limitations of the practice for mechanical meibomian gland expression (MMGE) were pain caused by forced evacuation of the gland, difficulty with adequate sustained temperature at the eyelid at therapeutic levels ≥ 40°C28, and duration of effect demonstrated in only one month. In the patients five sessions per year of this combined treatment for moderate and severe DGM was performet.

The aim of this study is to compare the safety and efficacy of one-session eyelid treatment with the ILux® DGM treatment device versus five sessions in MMGE consultation in patients with moderate and severe DGM in a follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years
* A history of self-reported dry eye symptoms for two months prior to study enrollment,
* Diagnosis of MGD Low delivery type, with mechanism obstructive and non- cicatricial with scores as follows: Ocular Surface Disease Index (OSDI) questionnaire ≥ 13, Non-Invasive Tear break-up time (NIBUT) lower than 10 seconds (The Sirius anterior segment analyzer (CSO, Florence, Italy).
* Meibomian gland scores (MGS) lower than 15.

Exclusion Criteria:

* A history of ocular surgery
* Allergic conjunctivitis
* Seborrheic dermatitis
* Rosacea
* Psoriasis
* Punctal plugs or previous punctal cautery
* Anterior or demodex blepharitis
* Cicatricial lid margin disease
* Ocular injury or trauma
* Chemical burns
* Limbal stem cell deficiency
* Active ocular infection or non-dry eye inflammation
* Aqueous-deficient dry eye
* Irregular cornea
* Lid abnormalities and systemic disease conditions
* Medications that cause dry eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Effectiveness defined as changes from baseline to 1, 3, 6, 9 and 12 months in Non Invasive Tear break-up time (NI-TBUT) in seconds. | 1 year
  NIBUT measured by SIRIUS device in seconds.
Effectiveness defined as changes from baseline to 1, 3, 6, 9 and 12 months in Meibomian gland scores (MGS). | 1 year
  Using a Meibomian Gland Evaluator (MGE 1000) to grade a total score for 15 meibomian glands in the lower eyelid evaluated in 3 areas: nasal (5 glands), medial (5 glands), and temporal (5 glands) expressed & graded from 0 to 3 (0 = no secretion, 1 = inspissated, 2 = cloudy, 3 = clear liquid).

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica de Oftalmología de Cali S.A, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: In 3 months
Access Criteria: Restricted access by request
URL: https://www.visionsana.com/